CLINICAL TRIAL: NCT06235112
Title: AI Detection of Incidental Coronary Artery Calcium to Enhance Cardiovascular Disease Prevention: A Multicenter Randomized Trial
Brief Title: AI Detection of Incidental Coronary Artery Calcium to Enhance Cardiovascular Disease Prevention
Acronym: AI INFORM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Nano-X Imaging Limited (Unknown)
Responsible Party: Principal Investigator, Daniel Michael Huck, MD, MPH, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023P002954
Record Dates: First submitted 2024-01-10; First posted 2024-01-31 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of two arms, involving notification to providers (vs non-notification)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Notification of Coronary Artery Calcification (Experimental): Notification to providers of the presence of coronary artery calcification automatically detected by AI based device (software) on chest CT.
  Recommendation of preventive therapy.
  Interventions: Device: Electronic health record-based notification of Nanox.AI Coronary Artery Calcification Assessment
- Non-notification of Coronary Artery Calcification (No Intervention): No notification to providers of the presence of coronary artery calcification on chest CT automatically detected by AI based device (software) on chest CT.
  No recommendation of preventive therapy.

INTERVENTIONS:
Device: Electronic health record-based notification of Nanox.AI Coronary Artery Calcification Assessment — The intervention involves electronic health record, email, or letter notification about the presence of coronary artery calcification on chest CT and recommendation of preventive therapy. This is based on results of the automatic detection of coronary artery calcification from AI device (software).
  Arms: Notification of Coronary Artery Calcification

SUMMARY:
AI INFORM is a multicenter randomized trial that will test the hypothesis that providing clinicians information on the presence and amount of coronary artery calcifications (CAC), will result in initiation or intensification of preventive therapies. The study will use a cloud-based artificial intelligence (AI) platform (Nanox.AI) that can analyze non contrast chest CT and estimate the amount of CAC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 40-75 with prior chest CT within last 3 years

Exclusion Criteria:

* Prior coronary artery disease
* Prior cancer
* Other life-limiting condition

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with initiation or intensification of lipid-lowering therapy after intervention | 6 months
  Initiation or intensification of therapy (yes/no) by 6 months after the intervention. Initiation: starting lipid-lowering therapy; intensification: increasing the dose of lipid-lowering therapy

SECONDARY OUTCOMES:
Average change in LDL-C after intervention | 12 months
  Average quantitative change in LDL-C (low-density lipoprotein cholesterol) between baseline and 12 months after intervention
Proportion of participants with downstream invasive or noninvasive testing after intervention | 12 months
  Composite outcome: Downstream testing (yes/no) including coronary artery calcium score, coronary CT angiography, invasive coronary angiography, or stress testing by 12 months after the intervention.
Proportion of participants with major adverse cardiovascular events after intervention | 12 months
  Composite outcome: Occurrence of an adverse cardiovascular event (yes/no) including cardiovascular death, myocardial infarction, or stroke by 12 months after the intervention
Proportion of participants with initiation or intensification of other preventive therapies after intervention | 6 months
  Initiation or intensification of preventive therapy (yes/no) by 6 months after the intervention. Preventive therapy includes any of the following: aspirin, antihypertensive therapy, metabolic therapy. Initiation: starting preventive therapy; intensification: increasing the dose of preventive therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared